CLINICAL TRIAL: NCT03742258
Title: A Phase 1 Study of R-CHOP Plus SYK Inhibitor TAK-659 for the Front-Line Treatment of High-Risk Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: Combination Chemotherapy and TAK-659 as Front-Line Treatment in Treating Patients With High-Risk Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 18H02; STU00207880 (CTRP (Clinical Trial Reporting Program)); NU 18H02 (Other: Northwestern University); P30CA060553 (NIH); NCI-2018-01917 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma Activated B-Cell Type; Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma, Not Otherwise Specified; T-Cell/Histiocyte-Rich Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; TAK-659; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- TAK-659 60mg + R-CHOP (Experimental): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV over 3-5 minutes, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning in cycle 2, patients also receive spleen tyrosine kinase inhibitor TAK-659 Dose Level 1 PO QD on days 1-21. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Biological: Rituximab; Drug: Spleen Tyrosine Kinase Inhibitor TAK-659; Drug: Vincristine Sulfate
- TAK-659 80mg + R-CHOP (Experimental): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV over 3-5 minutes, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning in cycle 2, patients also receive spleen tyrosine kinase inhibitor TAK-659 Dose Level 2 PO QD on days 1-21. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Biological: Rituximab; Drug: Spleen Tyrosine Kinase Inhibitor TAK-659; Drug: Vincristine Sulfate
- TAK-659 100mg + R-CHOP (Experimental): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV over 3-5 minutes, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning in cycle 2, patients also receive spleen tyrosine kinase inhibitor TAK-659 Dose Level 3 PO QD on days 1-21. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Biological: Rituximab; Drug: Spleen Tyrosine Kinase Inhibitor TAK-659; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Spleen Tyrosine Kinase Inhibitor TAK-659 — Given PO
  Other Names: Spleen Tyrosine Kinase Inhibitor TAK659; syk Inhibitor TAK-659; syk Inhibitor TAK659; syk-Inhibitor TAK-659; syk-Inhibitor TAK659; TAK-659; TAK659
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
The purpose of this research study is to evaluate a new investigational drug, TAK-659, given in combination with standard chemotherapy, for the treatment of Diffuse Large B-cell Lymphoma (DLBCL). ?Investigational? means that TAK-659 has not been approved by the United States Food and Drug Administration (FDA) for use as a prescription or over-the-counter medication to treat a certain condition. The primary purpose of this study is to find the appropriate and safe dose of the study drug to be used in combination with standard chemotherapy for the treatment of your disease and to determine how well the drug works in treating the disease. Other objectives include measuring the amount of the study drug in the body at different times after taking the study drug.

Participation in the study is expected to last for up to 3 years after receiving the last dose of the study drug. Patients will receive the study treatment for up to 18 weeks, as long as they are benefitting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability, and maximum tolerated dose of TAK-659 when combined with R-CHOP in the front-line treatment of high-risk diffuse large B cell lymphoma (DLBCL).

SECONDARY OBJECTIVES:

I. To assess preliminary efficacy of TAK-659 combined with R-CHOP in the front-line treatment of high-risk DLBCL.

EXPLORATORY OBJECTIVES:

I. To characterize the pharmacokinetics (PK) of TAK-659 in combination with R-CHOP.

OUTLINE: This is a dose-escalation study of spleen tyrosine kinase inhibitor TAK-659.

Patients receive rituximab intravenously (IV), cyclophosphamide IV, doxorubicin hydrochloride IV over 3-5 minutes, and vincristine sulfate IV on day 1, and prednisone orally (PO) on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning in course 2, patients also receive spleen tyrosine kinase inhibitor TAK-659 PO once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed diagnosis of DLBCL (including DLBCL not otherwise specified [NOS], DLBCL germinal center B-cell [GCB] type, DLBCL activated B cell [ABC]/non-GCB type, T cell/histiocyte-rich large B cell lymphoma, high-grade B cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, and high-grade B cell lymphoma NOS). NOTE: DLBCL transformed from low-grade lymphoma among treatment-naive patients or patients previously treated with a non-anthracycline containing regimen are permitted
* Patients may have completed the first cycle of R-CHOP (off study not combined with TAK-659) =< 21 days prior to the first dose of TAK-659 or plan to receive the first cycle of R-CHOP after registration
* Patients must have at least one high-risk feature, including:

  * ABC/non-GCB subtype determined by gene expression profiling or Hans algorithm by immunohistochemistry per treating institution standards
  * High-intermediate or high-risk group by National Comprehensive Cancer Network - International Prognostic Index (NCCN-IPI) with score >= 4, at time of diagnosis
  * MYC gene rearrangement (by [fluorescent in situ hybridization] FISH)
  * MYC overexpression by immunohistochemistry (IHC) (>= 40%) and BLC2 overexpression by IHC (>= 50%) or
  * Previously treated transformed low-grade lymphoma to large B cell lymphoma with prior treatment not including an anthracycline
  * NOTE: BCL2 and/or BCL6 aberrancy are not required for enrollment, but assessment for rearrangement by FISH and overexpression by IHC are required if there is presence of MYC rearranged by FISH
* Patients must have measurable disease (defined as >= 1.5 cm in diameter) with correlated fluorodeoxyglucose (FDG)-avidity on positron emission tomography (PET) scan with Deauville score of 4 or 5 at time of diagnosis
* Patients must have recovered (i.e., =< grade 1 toxicity) from the reversible effects of prior anticancer therapy, if applicable
* Life expectancy of greater than 3 months
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count >= 1000/mcL (within 14 days prior to registration)
* Platelets >= 75,000/mcl (NOTE: Patients with bone marrow involvement may be eligible with platelets >= 50,000) (within 14 days prior to registration)
* Hemoglobin >= 8 g/dL (within 14 days prior to registration)

  * NOTE: Red blood cell (RBC) and platelet transfusion allowed >= 14 days prior to registration
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN (within 14 days prior to registration)
* Creatinine clearance >= 60 mL/min either as estimated by the Cockcroft-Gault equation or based on urine collection (12 or 24 hours) (within 14 days prior to registration)
* Lipase =< 1.5 x ULN with no clinical symptoms suggestive of pancreatitis or cholecystitis (within 14 days prior to registration)
* Amylase =< 1.5 x ULN with no clinical symptoms suggestive of pancreatitis or cholecystitis (within 14 days prior to registration)
* Patients must have blood pressure =< grade 1

  * NOTE: Hypertensive patients are permitted if their blood pressure is controlled to =< grade 1 by hypertensive medications
* Female patients must meet at least one of the following criteria:

  * Are postmenopausal with last menstrual period at least 1 year before registration OR
  * Are surgically sterile, OR
  * If they are of childbearing potential

    * Agree to practice 1 highly effective method of contraception and one additional effective (barrier) method at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, or
    * Agree to practice true abstinence, when is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together
    * Agree not to donate eggs (ova) during the course of this study or 180 days after receiving their last dose of study drug
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 180 days after the last dose of study drug, or
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception. Female and male condoms should not be used together.)
  * Agree not to donate sperm during the course of this study or within 180 days after receiving their last dose of study drug
* Female of childbearing potential (FOCBP) must have a negative pregnancy test =< 7 days prior to registration on study
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Patients must have the ability to swallow oral medication
* Patients must be willing and able to complete study-required procedures

Exclusion Criteria:

* Patients with exposure to chemotherapy or immunotherapy =< 30 days prior to starting study treatment are not eligible

  * NOTE: Patients may receive at most 1 cycle of R-CHOP, rituximab, or systemic corticosteroids within this timeframe
  * NOTE: If patient is registered prior to completion of washout, start date of treatment will need to be confirmed prior to registration
* Patients with prior exposure to a SYK inhibitor are not eligible

  * NOTE: Examples of SYK inhibitors include fostamatinib (R788), entospletinib (GS-9973), cerdulatinib (PRT062070), and TAK-659
* Patients with untreated brain metastases or leptomeningeal metastases are not eligible
* Patients with known hypersensitivity (e.g. anaphylactic and anaphylactoid reactions) to TAK-659 or components of R-CHOP are not eligible
* Patients with history of drug-induced pneumonitis requiring treatment with steroids; history of idiopathic pulmonary fibrosis, organizing pneumonia, or evidence of active pneumonitis on screening imaging are not eligible

  * NOTE: A history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with known hepatitis B surface antigen positive, or known or suspected active hepatitis C infection are not eligible
* Patients who are known to be human immunodeficiency virus (HIV) positive are not eligible
* Patients must not have had autologous stem cell transplant within 6 months prior to registration
* Patients must have not had allogeneic stem cell transplant at any time
* Patients who have received systemic anticancer treatment (including investigational agents) or radiotherapy less than 3 weeks before the first dose of study treatment (=< 5 times half-life for large molecule agents or =< 4 weeks with evidence of disease progression if 5 times half-life is > 4 weeks) are not eligible

  * NOTE: Patients may receive R-CHOP cycle 1
  * NOTE: If patient is registered prior to completion of washout, start date of treatment will need to be confirmed prior to registration
* Use or consumption of the following substances is not permitted:

  * Medications or supplements that are known to be inhibitors of P-gp and/or strong reversible inhibitors of CYP3A within 5 times the inhibitor half-life (if a reasonable half-life estimate is known), or within 7 days (if a reasonable half-life estimate is unknown), before the first dose of study drug. The use of these agents is not permitted during the study
  * Medications or supplements that are known to be strong CYP3A mechanism-based inhibitors or strong CYP3A inducers and/or P-gp inducers within 7 days, or within 5 times the inhibitor or inducer half-life (whichever is longer), before the first dose of study drug. The use of these agents is not permitted during the study
  * Grapefruit-containing food or beverages within 5 days before the first dose of study drug. Note that grapefruit-containing food and beverages are prohibited during the study
* Patients who have major surgery, per principal investigator (PI) discretion, =< 14 days before the first dose of study drug and those who have not recovered fully from any complications from surgery are not eligible
* Patients who have systemic infection requiring parenteral antibiotic therapy or other serious infection (bacterial, fungal or viral) =< 21 days before the first dose of study drug are not eligible

  * NOTE: Patients who are at substantial risk of developing an infection may receive prophylaxis at the start of study treatment per investigator?s discretion
* Patients with an active secondary malignancy that requires treatment are not eligible

  * NOTE: Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection and are considered disease-free at the time of registration
* Patients with known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-659 are not eligible (this may include difficulty swallowing tablets or diarrhea > grade 1 despite supportive therapy)
* Patients who received treatment with high-dose corticosteroids for anticancer purposes =< 7 days before the first dose of TAK-659 are not eligible

  * NOTE: Prednisone and other steroids given as part of the R-CHOP regimen and as pre-medications are exceptions throughout the study. Patients may also receive steroids prior to starting chemotherapy to improve performance status. In other contexts, daily dose equivalent to 10 mg oral prednisone or less is permitted. Corticosteroids for topical use or in nasal spray or inhalers are allowed
* Patients who have known central nervous system (CNS) lymphomatous involvement are not eligible
* Patients who have an uncontrolled intercurrent illness, in the opinion of the investigator, including, but not limited to any of the following, are not eligible:

  * Uncontrolled pulmonary disease
  * Active CNS disease that would interfere with study participation
  * Active infection requiring parenteral systemic treatment
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient?s safety or study endpoints
* Patients with any of the following cardiovascular conditions are excluded:

  * Acute myocardial infarction within 6 months before starting study drug
  * Current or history of New York Heart Association class III or IV heart failure
  * Evidence of current, uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  * Fridericia corrected QT interval (QTcF) > 450 milliseconds (msec) (men) or > 475 msec (women) on a 12-lead electrocardiography (ECG) during the screening period
  * Abnormalities on 12-lead ECG including, but not limited to, changes in rhythm and intervals that, in the opinion of the investigator, are considered to be clinically significant
  * Abnormal left ventricular function (ejection fraction [EF] < 50%, as indicated by baseline echocardiography [ECHO])
* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on day 1 before first dose of TAK-659

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reem Karmali, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Cycle 1: R-CHOP
Arm/Group | TAK-659 60mg + R-CHOP | TAK-659 80mg + R-CHOP | TAK-659 100mg + R-CHOP
Started | 3 | 3 | 6
Completed | 3 | 3 | 6
Not Completed | 0 | 0 | 0
Period: Reached 1st Response Assessment
Arm/Group | TAK-659 60mg + R-CHOP | TAK-659 80mg + R-CHOP | TAK-659 100mg + R-CHOP
Started | 3 | 3 | 6
Cycle 2 | 3 | 3 | 6
Cycle 3 | 3 | 3 | 6
Reached 1st Response | 3 | 3 | 6
Completed | 3 | 3 | 6
Not Completed | 0 | 0 | 0
Period: Continued Treatment After 1st Response
Arm/Group | TAK-659 60mg + R-CHOP | TAK-659 80mg + R-CHOP | TAK-659 100mg + R-CHOP
Started | 3 | 3 | 6
Went on to Cycle 4 to End of Treatment | 3 | 3 | 6
Completed | 3 | 2 | 4
Not Completed | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Survival Follow-Up
Arm/Group | TAK-659 60mg + R-CHOP | TAK-659 80mg + R-CHOP | TAK-659 100mg + R-CHOP
Started | 3 | 3 (All patients who were treated with the study agent are followed for survival.) | 6 (All patients who were treated with the study agent are followed for survival.)
Completed | 3 | 3 | 4
Not Completed | 0 | 0 | 2
Not completed — Still in Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- TAK-659 80mg + R-CHOP; TAK-659 100mg + R-CHOP: Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV over 3-5 minutes, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning in cycle 2, patients also receive spleen tyrosine kinase inhibitor TAK-659 Dose Level 1 PO QD on days 1-21. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | TAK-659 60mg + R-CHOP | TAK-659 80mg + R-CHOP | TAK-659 100mg + R-CHOP | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 0 | 1 | 0 | 1
  30-39 | 0 | 0 | 0 | 0
  40-49 | 1 | 0 | 0 | 1
  50-59 | 1 | 0 | 2 | 3
  60-69 | 1 | 0 | 2 | 3
  70+ | 0 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 7
  Male | 2 | 1 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 3 | 1 | 4 | 8
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 3 | 5 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Determine the safety and establish the maximum tolerated dose of TAK-659 when combined with R-CHOP in the front-line treatment of high-risk DLBCL using only patients who are evaluable for dose limiting (DLT) toxicities. MTD for TAK-659 will be determined using a 3+3 dose escalation method. The starting dose was 60 mg with possible escalation to 80 mg and 100 mg. Patients may be de-escalated to 40 mg if DLT's were met at dose level 1.
Time Frame: The first 21 days after the participant received their first dose of TAK-695
Measure: Number; unit: mg TAK-659
Groups:
- Treatment (R-CHOP, TAK-659): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV over 3-5 minutes, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning in course 2, patients also receive spleen tyrosine kinase inhibitor TAK-659 PO QD on days 1-21. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  Cyclophosphamide: Given IV
  Doxorubicin Hydrochloride: Given IV
  Prednisone: Given PO
  Rituximab: Given IV
  Spleen Tyrosine Kinase Inhibitor TAK-659: Given PO
  Vincristine Sulfate: Given IV
Arm/Group | Treatment (R-CHOP, TAK-659)
Number analyzed (Participants) | 12
mg TAK-659 | 100

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Using Lugano criteria (2014), ORR will be defined as the percentage of subjects with a confirmed complete response (CR) or partial response (PR) as assessed by the investigators. Response will be assessed by positron emission tomography (PET)/computed tomography (CT).
Time Frame: PET/CT after the completion of Cycle 3
Population: The analysis population for this endpoint was defined in the protocol as all patients who completed 1 dose of TAK-659 and had 1 post-baseline disease assessment. Therefore, all 12 patients were analyzed as 1 group irrespective of the dose of TAK-659 they received.
Measure: Count of Participants; unit: Participants
Groups:
- TAK-659+ R-CHOP: Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV over 3-5 minutes, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Beginning in course 2, patients also receive spleen tyrosine kinase inhibitor TAK-659 PO QD on days 1-21. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  Cyclophosphamide: Given IV
  Doxorubicin Hydrochloride: Given IV
  Prednisone: Given PO
  Rituximab: Given IV
  Spleen Tyrosine Kinase Inhibitor TAK-659: Given PO
  Vincristine Sulfate: Given IV
Arm/Group | TAK-659+ R-CHOP
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS will be assessed using Kaplan-Meier curves at 12 month and 18 months during survival follow-up.
Time Frame: Up to 18 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of progression free survival
Arm/Group | Treatment (R-CHOP, TAK-659)
Number analyzed (Participants) | 12
percentage of progression free survival
  At 12 Months | .825 [.631 to 1]
  At 18 Months | .733 [.515 to 1]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 2 year period. Each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 30 days post last treatment.
Arm/Group | TAK-659 60mg + R-CHOP | TAK-659 80mg + R-CHOP | TAK-659 100mg + R-CHOP
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 6/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-659 60mg + R-CHOP (N=3) | TAK-659 80mg + R-CHOP (N=3) | TAK-659 100mg + R-CHOP (N=6)
Lung infection (Infections and infestations) | 0 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Bacteremia (Infections and infestations) | 0 | 0 | 2
Endocarditis infective (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 4
Thrush (Infections and infestations) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-659 60mg + R-CHOP (N=3) | TAK-659 80mg + R-CHOP (N=3) | TAK-659 100mg + R-CHOP (N=6)
Anemia (Blood and lymphatic system disorders) | 3 | 3 | 6
Eye disorders - Other, specify (Eye disorders) | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 3 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 5
Chills (General disorders) | 1 | 2 | 3
Edema face (General disorders) | 1 | 2 | 2
Fatigue (General disorders) | 2 | 2 | 6
Non-cardiac chest pain (General disorders) | 2 | 1 | 1
Pain (General disorders) | 1 | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 3 | 6
Alkaline phosphatase increased (Investigations) | 2 | 3 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 6
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 | 3 | 6
Creatinine increased (Investigations) | 1 | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 | 2 | 6
Lymphocyte count decreased (Investigations) | 3 | 3 | 6
Neutrophil count decreased (Investigations) | 1 | 1 | 5
Serum amylase increased (Investigations) | 1 | 2 | 5
Weight loss (Investigations) | 1 | 1 | 2
White blood cell decreased (Investigations) | 3 | 2 | 5
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 5
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 6
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Concentration impairment (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 3
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Hypertension (Vascular disorders) | 3 | 3 | 6
Palpitations (Cardiac disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 5
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 3
Floaters (Eye disorders) | 0 | 1 | 0
Periorbital edema (Eye disorders) | 0 | 1 | 2
Retinal vascular disorder (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 5
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Facial pain (General disorders) | 0 | 1 | 0
Fever (General disorders) | 0 | 2 | 3
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 0
Bacteremia (Infections and infestations) | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Cardiac troponin I increased (Investigations) | 0 | 1 | 3
GGT increased (Investigations) | 0 | 1 | 3
Lipase increased (Investigations) | 0 | 1 | 6
Lymphocyte count increased (Investigations) | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 1 | 5
Weight gain (Investigations) | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 4
Paresthesia (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 4
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 4
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 3
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Edema limbs (General disorders) | 0 | 0 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 5
Malaise (General disorders) | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Thrush (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 2
INR increased (Investigations) | 0 | 0 | 3
Investigations - Other, specify (Investigations) | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 0 | 4
Proteinuria (Renal and urinary disorders) | 0 | 0 | 4
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT03742258/Prot_SAP_000.pdf